CLINICAL TRIAL: NCT03523416
Title: Early Feasibility Study Of the Edwards APTURE Transcatheter Shunt System (ALT-FLOW US)
Brief Title: Early Feasibility Study - Edwards APTURE Transcatheter Shunt System
Acronym: ALT-FLOW US
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-02
Record Dates: First submitted 2018-04-12; First posted 2018-05-14 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Edwards Transcatheter Atrial Shunt System (Experimental)
  Interventions: Device: Transcatheter Atrial Shunt System

INTERVENTIONS:
Device: Transcatheter Atrial Shunt System — Transcatheter treatment of symptomatic left heart failure patients

SUMMARY:
The purpose of this study is to evaluate initial clinical safety, device functionality and effectiveness of the Edwards Transcatheter Atrial Shunt System.

DETAILED DESCRIPTION:
The early feasibility study of the Edwards Transcatheter Atrial Shunt System is a multi-center, prospective, early feasibility study to evaluate initial clinical safety, device functionality, and effectiveness of the Edwards Transcatheter Atrial Shunt System.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Heart Failure (HF):

  * NYHA class II with a history of > II; III; or ambulatory IV AND
  * ≥ 1 HF hospital admission; or treatment with IV or oral diuresis within 12 months; OR an NT-pro BNP value > 150 pg./ml in normal sinus rhythm, > 450 pg./ml in atrial fibrillation, or a BNP value > 50 pg./ml in normal sinus rhythm, > 150 pg./ml in atrial fibrillation within the past 6 months prior to study entry.
* On stable Guideline Directed Medical Therapy (GDMT) for heart failure
* At rest: elevated LAP (or PCWP) of > 15 mmHg and LAP (or PCWP) exceeds right atrial pressure (RAP) by > 5 mmHg AND/OR supine ergometer exercise, elevated LA (or PCWP) pressure of > 25 mmHg and LA (or PCWP) exceeds right atrial pressure (RAP) by > 10 mmHg
* Left Ventricular Ejection Fraction (LVEF) ≤ 40%
* Pulmonary Vascular Resistance (PVR) < 4.0 WU

Exclusion Criteria:

* Severe HF:

  * Stage D, non-ambulatory NYHA Class IV, transplant list
  * If BMI < 30, Cardiac index < 2.0 L/min/m2
  * If BMI ≥ 30, cardiac index < 1.8 L/min/m2
  * Left Ventricular End-Diastolic Diameter (LVEDD) > 8 cm
  * LVEF < 20%
* Valve disease: MR > 3+ or > moderate MS, TR > 2+, AR > 2+ or > moderate AS
* MI or therapeutic invasive cardiac procedure < 3 months
* TIA, stroke, CRT implanted < 6 months
* RV dysfunction > mild by TTE OR TAPSE < 1.2 OR RV size ≥ LV size by TTE, OR right ventricular fractional area change (RVFAC) ≤ 25%
* Dialysis OR renal dysfunction (S-CR > 2.5 mg/dl OR eGFR < 25 ml/min/1.73m2)
* 6MWT < 50m OR > 600m
* Active endocarditis or infection < 3 months
* Mean Right Atrial Pressure (mRAP) > 15 mmHg at rest
* Body Mass Index (BMI) ≥ 45 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Rate of major cardiac/cerebrovascular/renal events and re-intervention (Safety Endpoint) | 30 days
  Composite of major adverse cardiac, cerebrovascular, renal events (MACCRE) and re-intervention for study device related complications at 30 days.

SECONDARY OUTCOMES:
Rate at which device is successfully implanted (Device Success) | Day 0
  Device is deployed as intended and the delivery system is successfully removed as intended at the time of the patient's exit from the implant procedure room.
Rate at which device is patent and subject is discharged from hospital without the need for additional intervention for the device (Procedural Success) | 10 days post-op
  Device success with evidence of shunt patency and hospital discharge without the need for additional surgical or percutaneous intervention related to the study device including unacceptable Qp/Qs values.
Rate at which the procedure is successful without major cardiac/cerebrovascular/renal events and re-intervention (Clinical Success) | 30 days
  Procedural success without major adverse cardiac, cerebrovascular, and renal events (MACCRE) and re-intervention for study device related complications at 30 days.
Change in the ratio of systemic blood flow (Qs) to the pulmonary blood flow (Qp), called "Qp/Qs", from Baseline to Follow Up | 3 months, 6 months
  Change in Qp/Qs value from Baseline to Follow Up (3Month, 6Month)
Change in pulmonary capillary wedge pressure (PCWP) from Baseline to Follow Up | 3 months, 6 months
  Change in PCWP value from Baseline to Follow Up (3Month, 6Month)
Change in mean systolic & diastolic pulmonary artery pressure (PAP) and change in mean right atrial pressure (RAP) from Baseline to Follow Up | 3 months, 6 months
  Change in PAP and RAP values from Baseline to Follow Up (3Month, 6Month) under the same test conditions (e.g. comparison in the value at rest at baseline, to at rest at follow up; comparison in the value at exercise at baseline, to at exercise at follow up)
Change in Pulmonary Vascular Resistance (PVR) from Baseline to Follow Up | 3 months, 6 months
  Change in PVR value from Baseline to Follow Up (3Month, 6Month) under the same test conditions (e.g. comparison in the value at rest at baseline, to at rest at follow up; comparison in the value at exercise at baseline, to at exercise at follow up)
Change in two parameters related to Tricuspid Annular Plane Excursion (TAPSE) from Baseline to Follow Up | 3 months, 6 months
  Change in two parameters from Baseline to Follow Up (3Month, 6Month): 1. "TAPSE", Tricuspid Annular Plane Excursion 2. "TAPSE/sPAP", Tricuspid Annular Plane Excursion (TAPSE) divided by the systolic pulmonary Artery Pressure (sPAP)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - UC San Diego Health, La Jolla, California
  - University California San Francisco, San Francisco, California
  - University of Florida Health - Jacksonville, Jacksonville, Florida
  - St. Vincent Medical Group, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Abbott Northwestern, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Montefiore Medical Center, The Bronx, New York
  - Atrium Health, Charlotte, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Fioretti F, Hibbert B, Eckman PM, Simard T, Labinaz M, Nazer B, Wiley M, Gupta B, Sauer AJ, Shah H, Sorajja P, Pineda AM, Missov E, Aldaia L, Koulogiannis K, Gray WA, Zahr F, Butler J. Left Atrial-to-Coronary Sinus Shunting in Heart Failure With Mildly Reduced or Preserved Ejection Fraction: The ALT-FLOW Trial (Early Feasibility Study) 2-Year Results. JACC Heart Fail. 2025 Jun;13(6):987-999. doi: 10.1016/j.jchf.2025.02.003. Epub 2025 Feb 11. PMID 40019407